CLINICAL TRIAL: NCT02821247
Title: A Prospective obsERvational Study to asSEss the Effectiveness of Intravitreal Aflibercept Injection in roUtine Clinical Practice in Treatment Naive patientS With Wet Age-related Macular Degeneration in Greece
Brief Title: Prospective Observational Study to Assess Effectiveness of Intravitreal Aflibercept in Patients With Wet Macular Degeneration in Greece
Acronym: PERSEUS-GR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18033; SIRIUS/OS-CY-1668 (Other: company internal)
Record Dates: First submitted 2016-05-11; First posted 2016-07-01 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Choroidal Neovascularization; Macular Degeneration
Keywords: Treatment Naïve Patients
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Aflibercept: Adult wet Age Related Macular degeneration (AMD) treatment naïve partcipants were treated with intravitreal aflibercept injection
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Intravitreal injection; should comply with the recommendations written in the local Summary of Product Characteristics (SPC) of the product
  Other Names: VEGF Trap-Eye

SUMMARY:
This is a prospective, observational, multi-center, study. The study will be conducted in approximately 12 ophthalmological clinics and practices throughout Greece. It is planned to collect data on treatment of wet Age related Macular Degeneration (wAMD) from about 120 patients for which the decision to treat with intravitreal aflibercept injections is made at the discretion of the attending physician, according to his/her medical practice. Visits will be performed at baseline, aflibercept first injection (if different from enrollment) and at 12 and 24 months. The 12 and 24 month comprise the data collection visits during which any data generated in the period preceding these visits will be recorded.

All required information for the purposes of this study will be collected using electronic Case Record Form (eCRF). The web-based electronic data capture (EDC) application will be specifically designed for the needs of the study and will adhere to all applicable data protection regulations and requirements with regard to electronic records.

The study observation period for each patient enrolled in this study is the time from the beginning of treatment with intravitreal aflibercept injection up to two years or until discontinuation of intravitreal aflibercept injection-treatment due to any reason including withdrawal of consent or patient loss from follow-up.

DETAILED DESCRIPTION:
Rationale and background Age-related macular degeneration (AMD) is the most common degenerative disease of the macula and the most common cause of legal blindness in the Western world. AMD is a disease of the elderly affecting 10% of individuals aged 65 to 74 years and 30% of those aged 75 to 85 years. Two forms of AMD can be distinguished. The dry form is more benign accounting for 90% of all AMD cases, but only for 10% of cases of blindness due to AMD. On the other hand wet AMD affects only 10% of AMD patients. However, it is more aggressive and rapidly progresses. Wet AMD (wAMD) accounts for 80% of cases of severe visual impairment and represents the majority of cases of legal blindness. Thus, wet or neovascular AMD is a disease with a great impact on both visual acuity and patients' quality of life.

About 1% of the population is affected by wAMD between 65-74 years of age, 5% between 75-84 years of age and 13% in people 85+ years. Given that wAMD is a strongly age-dependent disease its prevalence is expected to significantly increase in western countries (including Greece) in the near future. Therefore, early diagnosis and proper treatment will be a major public health concern.

AMD is diagnosed by stereoscopic biomicroscopy and additional examinations of the macula, such as fluorescein angiography (FA), indocyanine green angiography (ICGA) and optical coherence tomography (OCT). The patient's visual status can be monitored with the Snellen chart and Early Treatment Diabetic Retinopathy Study (ETDRS) chart, the Snellen chart being most often used in Greece.

Wet AMD is caused by choroidal neovascularization (CNV) whereby new abnormal blood vessels spread beneath the retina. These vessels may rupture and cause retinal damage. In addition, vascular leakage may cause thickening and oedema of the retina, which is thought to contribute to vision loss. Vascular endothelial growth factor (VEGF) and placental growth factor (PlGF) play a pivotal role in this scenario. VEGF-A and PlGF are members of the VEGF family of angiogenic factors that act as potent mitogenic, chemotactic, and vascular permeability factors for endothelial cells. VEGF acts via two receptor tyrosine kinases-VEGFR-1 and VEGFR-2-which are located on the surface of endothelial cells. PlGF binds only to VEGFR-1, which is also present on the surface of leukocytes. Excessive activation of these receptors by VEGF-A can induce pathological neovascularization and excessive vascular permeability. PlGF can synergize with VEGF-A in these processes, and is also known to promote leukocyte infiltration and vascular inflammation.

Treatment paradigms for wet AMD have changed tremendously since anti-VEGF treatment (inhibition of all VEGF-A Isoforms) was introduced. As a consequence, most previous therapy approaches lost significance and are applied in rare cases only. The pan-anti-angiogenesis treatment with ranibizumab was the first to show significant improvements in visual acuity of patients suffering from wAMD, thus becoming the first-choice therapy for most patients. The phase III clinical trials MARINA and ANCHOR have shown that ranibizumab applied every month is highly effective in improving visual impairment. However, in addition to the small risk of endophthalmitis associated with intravitreal injections, monthly treatment, which may continue for a patient's lifetime, is extremely burdensome to patients, their caregivers, ophthalmologists and the healthcare system. As a consequence, in clinical practice the monthly treatment regimen of ranibizumab is often altered to less frequent dosing intervals to reduce the associated treatment burden, although this may result in notably reduced efficacy.

Results from observational studies such as WAVE and AURA, which investigated wAMD patients treated with Lucentis (ranibizumab) in a real life setting in western countries, suggest that these patients are not treated according to a continuous treatment pattern and are also undertreated resulting in suboptimal treatment effects. In the WAVE Study (n=2587) patients received 4.3 injections during the first treatment year and the visual acuity returned to the baseline visual acuity at the end of the year. In the AURA study (n=420), German cohort, patients received 4.3 injections in the first year and only 2.1 injections during the second year. The visual acuity declined during year 1 to -1.4 letters and further declined to -2.4 letters during year 2 compared to baseline. In the AURA study (n =365), Italian cohort, patients received 3.9 injections in the first year and only 1.4 injections during the second year. The visual acuity declined during year 1 to 0 letters and further declined to -2.9 letters during year 2 compared to baseline .

Intravitreal aflibercept is the next generation of anti-angiogenesis treatments which also introduces a new proactive every-other-month treatment regimen (after 3 monthly injections) in the first year, followed by individually extended treatment intervals afterwards. Aflibercept is a fusion protein consisting of portions of human VEGF receptors 1 and 2 extracellular domains fused to the Fc portion of human IgG1. It is purified and formulated as a solution for intravitreal use. As such, aflibercept acts as a soluble decoy receptor that binds VEGF-A and PlGF with higher affinity than naturally occurring VEGF receptors. Thus aflibercept competitively inhibits VEGF-A and PIGF binding to the cognate VEGF receptors and their activation.

Intravitreal aflibercept was recently approved by the European Medicines Agency (EMA) in November 2012. The aims of this study are to collect data on the effectiveness of intravitreal aflibercept and to evaluate follow-up as well as treatment patterns in treatment naive patients with wAMD in routine clinical practice in Greece treated with intravitreal aflibercept injection.

Research questions and objectives The main objectives of this observational study are to evaluate the effectiveness of intravitreal aflibercept injection and to describe routine clinical practice monitoring and treatment patterns in treatment-naïve wAMD patients in Greece.

Primary objective

The primary objective in this study is:

* To evaluate the effectiveness of intravitreal aflibercept injection by assessing the change in best corrected visual acuity (BCVA; defined as visual acuity with manifest refraction) from baseline at the 12-month timepoint, in treatment naive patients with wAMD in routine clinical practice in Greece.

Secondary objective(s)

The secondary objectives in this study are:

* To evaluate the effectiveness of intravitreal aflibercept injection by assessing the change in BCVA (with manifest refraction) from baseline at the 24-month timepoint
* To evaluate the effectiveness of intravitreal aflibercept injection by assessing the change in visual acuity with glasses from baseline to the 24-month timepoint
* To assess the change in central retinal thickness at 12 and 24 months
* To assess the proportion of patients with no fluid at 12 and 24 months
* To assess the disease activity monitoring patterns and the treatment patterns used in routine clinical practice (e.g. number of evaluation visits, injection visits, combined visits, OCT tests, visual acuity tests, fundoscopy tests, Fluorescein Angiography (FA) and Indocyanine Green Angiograpy (ICGA tests).

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive patients with wet AMD for whom the decision to be treated with intravitreal aflibercept injection in accordance with the Summary of Product Characteristics was made.
* Patients having signed the informed consent.

Exclusion Criteria:

* Contraindications as listed in the local Summary of Product Characteristics.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Any prior or concomitant therapy with any other agent (including among others, anti-VEGF agents and photodynamic therapy) to treat wet AMD in the study eye.
* Patients with previous exposure to systemic anti-VEGF treatment.
* Patients participating in an investigational program with interventions.
* Previous macular surgery, including laser, for any retinal pathology in the study eye.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients treated with Aphlibercept as first treatment for wAMD ( Treatment Naïve Patients).
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Mean change of visual acuity from baseline to 12 months | At baseline and 12 months

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) (with manifest refraction) from baseline at the 24-month timepoint | At baseline, At 24 months
Change in visual acuity with glasses from baseline to the 24-month timepoint | At baseline, At 24 months
Change in central retinal thickness (OCT measurement) at 12 and 24 months | At 12 months, At 24 months
Proportion of patients with no fluid at, 12 and 24 months | At 12 months, At 24 months
Total number of routine clinical evaluation (monitoring) visits at 12 and 24 months | At 12 months, At 24 months
Number of optical coherence tomography (OCT) assessments per patient | At 12 months, At 24 months
Number of visual acuity tests | At 12 months, At 24 months
Number of fundoscopy examinations | At 12 months, At 24 months
Total number of injection visits at 12 and 24 months | At 12 months, At 24 months
Number of combined visits (monitoring and injection) at 12 and 24 months | At 12 months, At 24 months
Number of fluorescein angiography (FA) tests / patient at 12 and 24 months | At 12 months, At 24 months
Number of indocyanine green angiography (ICGA) tests / patient at 12 and 24 months | At 12 months, At 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Greece